CLINICAL TRIAL: NCT00349752
Title: A Phase IIIb Multicenter, Double-blind, Placebo-controlled,Randomized Trial to Examine the Corticosteroid-sparing Effect of Certolizumab Pegol in Patients With Moderate to Severe Crohn's Disease.
Brief Title: Corticosteroid Sparing Effect of Certolizumab in Crohn's Disease
Acronym: COSPAR1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment was stopped early due to slow enrolment of this population. With no safety concerns, the study continued normally for subjects already recruited
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C87059; 2006-003870-88 (EudraCT Number)
Expanded Access: NCT03559660 (No longer available)
Record Dates: First submitted 2006-06-30; First posted 2006-07-10 (Estimated); Results first posted 2010-12-01 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2010-10

CONDITIONS: Crohn's Disease
Keywords: certolizumab pegol; Cimzia; Crohn's Disease; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Certolizumab pegol 400 mg (Experimental): Certolizumab pegol 400 mg
  Interventions: Biological: certolizumab pegol 400 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: certolizumab pegol 400 mg — Certolizumab pegol 400 mg provided in solution for subcutaneous injection (2 x 200 mg/mL) in single-use vials for administration at Weeks 0, 2, 4 and then every 4 weeks until Week 36. Two vials will be required for each dosing.
  Other Names: Cimzia; CDP870; CZP
  Arms: Certolizumab pegol 400 mg
Other: Placebo — Placebo (commercially available sodium chloride 0.9% (preservative free)) provided for subcutaneous injection in single-use vials for administration at Weeks 0, 2, 4 and then every 4 weeks until Week 36. Two vials will be required for each dosing.
  Arms: Placebo

SUMMARY:
The current study is designed to measure the corticosteroid-sparing effect of certolizumab pegol using a defined schedule of corticosteroid tapering in subjects with moderate to severe Crohn's disease. Subjects had to be in remission (CDAI<=150) and receiving corticosteroids at a dose no higher than 30 mg/day prednisone or equivalent during the week prior to randomization.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 18 years or older with moderate to severe Crohn's disease (Crohn's Disease Activity Index (CDAI) score of ≥ 220 ≤450)

Exclusion Criteria:

* Active or draining fistula present at screening
* Lactating and/or pregnant female subjects
* A history of any health condition that could potentially interfere with the disease and/or the treatment
* A history of an adverse reaction to polyethylene glycol (PEG) or a protein medicinal product
* Any other condition which in the Investigator's judgment would make the patient unsuitable for inclusion in the study
* History of drug or alcohol abuse in the prior year
* Receipt of any experimental therapy within or outside a clinical trial in the 3 months prior to Visit 0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2006-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (68):
- United States (54):
  - Birmingham, Alabama
  - Montgomery, Alabama
  - Tucson, Arizona
  - La Jolla, California
  - Oceanside, California
  - Orange, California
  - Palo Alto, California
  - Roseville, California
  - Golden, Colorado
  - Clearwater, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - North Miami Beach, Florida
  - Sarasota, Florida
  - Winter Park, Florida
  - Marietta, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Bloomington, Indiana
  - Topeka, Kansas
  - Bowling Green, Kentucky
  - Louisville, Kentucky
  - Metairie, Louisiana
  - Annapolis, Maryland
  - Newton, Massachusetts
  - Chesterfield, Michigan
  - Dearborn, Michigan
  - Troy, Michigan
  - Rochester, Minnesota
  - Ocean Springs, Mississippi
  - Kansas City, Missouri
  - Mexico, Missouri
  - New York, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Tulsa, Oklahoma
  - Columbia, South Carolina
  - Germantown, Tennessee
  - Austin, Texas
  - Irving, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Chesapeake, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
  - Monroe, Wisconsin
- Canada (9):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Abbotsford, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - London, Ontario
  - Toronto, Ontario
  - Saskatoon, Saskatchewan
- Germany (5):
  - Frankfurt
  - Heidleberg
  - Jena
  - Magdeburg
  - Ulm

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Randomized Trial to Examine the Corticosteroid-sparing Effect of Certolizumab Pegol in Subjects With Moderate to Severe Crohn's Disease from November 2006 to July 2009
Groups:
- Certolizumab Pegol 400 mg: Certolizumab pegol 400 mg provided in a solution for subcutaneous injection (2 x 200 mg/mL) in single-use vials for administration at Weeks 0, 2, 4 and then every 4 weeks until Week 36
- Placebo: Placebo provided for subcutaneous injection in 2 single-use vials for administration at Weeks 0, 2, 4 and then every 4 weeks until Week 36
Period: Overall Study
Arm/Group | Certolizumab Pegol 400 mg | Placebo
Started | 87 | 87
Completed | 28 | 23
Not Completed | 59 | 64
Not completed — Adverse Event | 8 | 12
Not completed — Lack of Efficacy | 37 | 42
Not completed — Lost to Follow-up | 4 | 2
Not completed — Personal reasons | 6 | 5
Not completed — Other: Required exclusionary medication | 0 | 1
Not completed — Other: Non compliance | 0 | 1
Not completed — Other: Patient stopped steroids | 0 | 1
Not completed — Other: Patient's steroid use | 1 | 0
Not completed — Other: Ineligible | 1 | 0
Not completed — Other: Inadvertently unblinded | 1 | 0
Not completed — Other:History of squamous cell carcinoma | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Certolizumab Pegol 400 mg | Placebo | Total
Number analyzed (Participants) | 87 | 87 | 174
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 85 | 170
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.77 (13.20) | 39.73 (13.31) | 40.25 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 45 | 97
  Male | 35 | 42 | 77
Region of Enrollment [Number; unit: participants]
  United States | 65 | 68 | 133
  Canada | 18 | 11 | 29
  Germany | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Have Been Withdrawn From Prednisone or Prednisolone Therapy According to the Corticosteroid Tapering Schedule and Have Remained Off Corticosteroids and in Disease Remission at Week 38
Description: The Crohn's Disease Activity Index (CDAI) is used to quantify the symptoms of subjects with Crohn's disease. A CDAI score of 150 or below indicates disease remission and a score above 450 indicates extremely severe disease.
Time Frame: Week 38
Population: Intention-to-treat (ITT) population which consists of all randomized subjects who received at least one injection of study medication. In the analyses of remission rates, subjects for whom it is impossible to assess the remission status will be conservatively considered as non-remitters in the calculations.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol 400 mg | Placebo
Number analyzed (Participants) | 87 | 87
percentage of subjects | 26.4 | 21.8

2. Secondary Outcome: Percentage of Subjects With Continuous Remission Off Steroids at Week 38
Description: The Crohn's Disease Activity Index (CDAI) is used to quantify the symptoms of subjects with Crohn's disease. A CDAI score of 150 or below indicates disease remission and a score above 450 indicates extremely severe disease. A subject with continuous remission off steroids at Week 38 is a subject in remission (CDAI =< 150) from the visit when he stops taking steroids to Week 38 and is off corticosteroids until Week 38.
Time Frame: Week 38
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol 400 mg | Placebo
Number analyzed (Participants) | 87 | 87
percentage of subjects | 16.1 | 14.9

3. Secondary Outcome: Cumulative Percentage of Subjects With Relapse/Treatment Failure at Week 38
Description: A subject with relapse/ treatment failure has a Crohn's Disease Activity Index (CDAI) > 150 and an increase in CDAI of >= 70 points versus Week 0. [The CDAI is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 or below indicates disease remission and a score above 450 indicates extremely severe disease.]
Time Frame: Week 38
Population: Of 87 (Placebo) and 87 (Certolizumab pegol 400 mg) subjects randomized, 85 and 87 subjects respectively are included in summary of Week 38, based on conditional intention-to-treat population, consisting of all randomized subjects who received at least one injection of study medication, excluding those who were not in remission (CDAI>150) at Week 0
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol 400 mg | Placebo
Number analyzed (Participants) | 87 | 85
percentage of subjects | 57.5 | 56.5

4. Secondary Outcome: Time to Relapse/Treatment Failure During the 38-week Double-blind Treatment Period
Description: as for outcome 3
Time Frame: During the 38-week double-blind treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Certolizumab Pegol 400 mg | Placebo
Number analyzed (Participants) | 87 | 85
days | 83.5 (61.8) | 81.9 (70.4)

5. Secondary Outcome: Per-subject Median Weekly Dose of Corticosteroids Over the 38-week Double-blind Treatment Period
Description: The median weekly dose of corticosteroids is calculated for each subject, and these per-subject median values are further summarized by treatment group. The mean of the per-subject median doses in each treatment group is presented here.
Time Frame: Over the 38-week double-blind treatment period
Population: 87 (Placebo) and 87 (Certolizumab pegol 400 mg) subjects randomized are included in the summary based on the intention-to-treat (ITT) population. Of the 87 subjects in the placebo group, 1 subject taking a daily dose of 3g with a rectal route has been excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mg per week
Arm/Group | Certolizumab Pegol 400 mg | Placebo
Number analyzed (Participants) | 87 | 86
mg per week | 88.66 (38.72) | 122.47 (210.15)

6. Secondary Outcome: Per-subject Cumulative Dose of Corticosteroids Over the 48-week Study Period
Description: The cumulative dose of corticosteroids over the 48-week study period is calculated for each subject individually. The mean of these values for each treatment group is presented here.
Time Frame: Over the 48-week study period
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Certolizumab Pegol 400 mg | Placebo
Number analyzed (Participants) | 87 | 86
mg | 792.68 (438.14) | 1294.96 (4459.27)

7. Secondary Outcome: Change From the 6-week run-in Period in Per-subject Median Weekly Dose of Corticosteroids Over the 38-week Double-blind Treatment Period
Description: The run in period lasted a minimum of 1 week and a maximum of 6 weeks. During this period subjects were treated with any dose or type of systemic corticosteroids the Investigator felt was appropriate. To be eligible for study randomization, subjects must have been in remission (CDAI ≤150 points) and receiving corticosteroids at a dose no higher than 30 mg/day prednisone or equivalent during the week prior to randomization. Subjects who did not meet these criteria were not randomized and were withdrawn from the study.
Time Frame: 6-week run-in period, 38-week double-blind treatment period
Population: Of the 87 (Placebo) and 87 (Certolizumab pegol 400 mg) subjects randomized, 86 in each group had available values at the 6-week run-in period and over the 38-week double-blind treatment period.
Measure: Mean (Standard Deviation); unit: mg per week
Arm/Group | Certolizumab Pegol 400 mg | Placebo
Number analyzed (Participants) | 86 | 86
mg per week | -111.20 (64.60) | -78.04 (202.55)

8. Secondary Outcome: Crohn's Disease Activity Index (CDAI) Score at Week 38
Description: The Crohn's Disease Activity Index (CDAI) is used to quantify the symptoms of subjects with Crohn's disease. A score of 150 or below indicates disease remission and a score above 450 indicates extremely severe disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Week 38
Population: Of the 87 (Placebo) and 87 (Certolizumab pegol 400 mg) subjects randomized, 22 and 27 subjects respectively are included in the summary of the Week 38, based on the intention-to-treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Certolizumab Pegol 400 mg | Placebo
Number analyzed (Participants) | 27 | 22
score on a scale | 78.90 (65.05) | 73.42 (61.09)

9. Secondary Outcome: Change From Baseline in CDAI Score at Week 38
Description: as for outcome 8
Time Frame: Week 0, Week 38
Population: Of the 87 (Placebo) and 87 (Certolizumab pegol 400 mg) subjects randomized, 22 and 27 subjects respectively had available values at Baseline and at Week 38 and are included in the summary based on the intention-to-treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Certolizumab Pegol 400 mg | Placebo
Number analyzed (Participants) | 27 | 22
score on a scale | -25.50 (53.48) | -18.36 (75.97)

10. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score at Week 38
Description: The total IBDQ score will be derived as the sum of the responses (each ranging from 1 to 7) to all 32 questions on the IBDQ and can therefore range from 32 to 224. A higher score indicates a better quality of life. IBDQ remission is defined as a subject having an IBDQ total score >= 170 points.
Time Frame: Week 38
Population: Of the 87 (Placebo) and 87 (Certolizumab pegol 400 mg) subjects randomized, 23 and 27 subjects respectively had available values at Week 38 and are included in the summary based on the intention-to-treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Certolizumab Pegol 400 mg | Placebo
Number analyzed (Participants) | 27 | 23
score on a scale | 174.7 (25.7) | 168.6 (23.4)

11. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score at Week 38
Description: The total IBDQ score will be derived as the sum of the responses (each ranging from 1 to 7) to all 32 questions on the IBDQ and can therefore range from 32 to 224. A higher scores indicates a better quality of life. IBDQ response is defined as an increase from baseline in the IBDQ total score >= 16 points.
Time Frame: Week 0, Week 38
Population: Of the 87 (Placebo) and 87 (Certolizumab Pegol 400 mg) subjects randomized, 23 and 26 subjects respectively had available values at Baseline and Week 38 and are included in the summary based on the intention-to-treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Certolizumab Pegol 400 mg | Placebo
Number analyzed (Participants) | 26 | 23
score on a scale | 12.6 (23.2) | 1.5 (21.5)

ADVERSE EVENTS:
Time Frame: 48-week study period
Arm/Group | Certolizumab Pegol 400 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 9/87 | 8/87
Other Adverse Events (participants affected / at risk) | 70/87 | 73/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol 400 mg (N=87) | Placebo (N=87)
Bundle Branch Block Left (Cardiac disorders) | 1 (1) | 0 (0)
Crohn's Disease (Gastrointestinal disorders) | 0 (0) | 5 (5)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic Stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileal Stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 2 (2) | 0 (0)
Granuloma (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abscess Intestinal (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Grand Mal Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol 400 mg (N=87) | Placebo (N=87)
Crohn's Disease (Gastrointestinal disorders) | 35 (35) | 39 (40)
Abdominal Pain (Gastrointestinal disorders) | 8 (10) | 11 (14)
Nausea (Gastrointestinal disorders) | 9 (9) | 8 (12)
Vomiting (Gastrointestinal disorders) | 10 (13) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 4 (5)
Abdominal Distension (Gastrointestinal disorders) | 7 (7) | 2 (4)
Abdominal Pain Lower (Gastrointestinal disorders) | 5 (5) | 4 (8)
Flatulence (Gastrointestinal disorders) | 3 (3) | 5 (5)
Fatigue (General disorders) | 8 (9) | 7 (9)
Pyrexia (General disorders) | 5 (6) | 7 (8)
Injection Site Reaction (General disorders) | 6 (9) | 1 (1)
Nasopharyngitis (Infections and infestations) | 12 (14) | 13 (15)
Urinary Tract Infection (Infections and infestations) | 7 (11) | 8 (10)
Sinusitis (Infections and infestations) | 5 (6) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (15) | 9 (10)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 9 (13) | 5 (5)
Headache (Nervous system disorders) | 19 (47) | 13 (23)
Haematuria (Renal and urinary disorders) | 5 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (6) | 6 (7)

LIMITATIONS AND CAVEATS:
Recruitment was stopped early due to slow enrolment of this population. With no safety concerns, the study continued normally for the 174 subjects already recruited. Results should be treated with caution due to the early termination of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.